CLINICAL TRIAL: NCT03911219
Title: Multicenter Study to Evaluate the Impact of eHealth Monitoring on Overall Survival in Patients With Metastatic Non-squamous NSCLC or Extensive-stage SCLC or Advanced TNBC Under First-line Treatment With Atezolizumab in Combination With Chemotherapy
Brief Title: Impact of eHealth Monitoring on Overall Survival in Patients With Metastatic NSCLC / Extensive-stage SCLC / Advanced TNBC Under First-line Treatment With Atezolizumab Plus Chemotherapy
Acronym: CHAPLIN
Status: Completed | Type: Observational
Sponsor: iOMEDICO AG (Industry)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Other Study IDs: iOM-100392; ML41161 (Other: Roche)
Record Dates: First submitted 2019-04-01; First posted 2019-04-11 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-10

CONDITIONS: Stage IV Non-small Cell Lung Cancer; Extensive-stage Small Cell Lung Cancer; Advanced (Locally Advanced and Inoperable or Metastatic), PD-L1 IC-positive TNBC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- CANKADO (Arm A): CANKADO application as eHealth support system: Patients use CANKADO for regular symptom self-reporting in addition to standard of care symptom management.
  Interventions: Other: eHealth system support for symptom management via CANKADO
- Control (Arm B): Control arm without eHealth support: Patients recieve standard of care symptom management.

INTERVENTIONS:
Other: eHealth system support for symptom management via CANKADO — Regular use of eHealth support system CANKADO by the patient: symptom self-reporting triggering alerts to the patient; in addition to standard of care symptom management.
  Groups: CANKADO (Arm A)

SUMMARY:
The current study is aimed to test the benefit of a web-based application tool in NSCLC, SCLC and TNBC patients during the recently approved first-line treatment strategy with atezolizumab in combination with chemotherapy.

DETAILED DESCRIPTION:
Checkpoint inhibitors represent new, promising treatment opportunities in the palliative lung cancer setting. Among programmed cell death-1 (PD-1) and programmed cell death ligand-1 (PD-L1) inhibitors, atezolizumab (Tecentriq® ), a PD-L1 inhibitor, has been shown to ameliorate outcomes for NSCLC patients with metastatic disease: The open-label phase II multicenter studies POPLAR and BIRCH revealed an improved overall response rate and a benefit in overall survival (OS) under atezolizumab monotherapy. The open-label, randomized phase III OAK trial led to atezolizumab approval as monotherapy for patients with metastatic NSCLC whose disease progressed during or following platinumcontaining chemotherapy regardless of PD-L1 status.

Despite these developments, platinum-based chemotherapy regimens are still standard of care for lung cancer without druggable alterations. Lately combining conventional chemotherapeutics with immunotherapy showed promising results: A phase I study of first-line atezolizumab plus chemotherapy demonstrated efficacy regardless of PD-L1 status and an acceptable safety profile in multiple tumor types. Accordingly, ongoing phase III trials address potential benefits of platinum-based immunotherapy combinations in comparison to standard platinum-containing regimens in first-line NSCLC and SCLC. If additional bevacizumab might further enhance atezolizumab efficacy by inhibiting vascular Endothelial Growth Factor (VEGF)-related immunosuppression is currently investigated in the IMpower150 trial.

Patients under intensive care for advanced cancers develop symptoms due to cancer progression and, possibly, due to therapy-related sideeffects. These symptoms are often not detected promptly by the treating physician leading to functional impairment and deconditioning of the patient's status with potential implications for the general outcome. Improved symptom control in late-stage cancer under exhaustive therapy regimens was achieved through intensified symptom management. Systematic collection of symptom information by electronic patientreported outcomes (ePROs) in addition to clinical routine provides an attractive basis for intensified symptom management. However, despite new, intriguing results, the proof of a significant benefit (defined as primary outcome measure) under first-line treatment is still limited in oncology trials.

In the palliative setting of lung cancer, routine treatment monitoring includes imaging at certain intervals. However, as approaching imaging assessments clarify the patient's fate, they are often a source for anxiety and concern. Additionally, patients with emerging symptoms often wait until the next routinely scheduled consultation with their treating oncologist. As a consequence, tumor progression without therapeutic hindrance over several weeks may occur and naturally shorten the patient's survival time. Clinical monitoring via self-assessed symptom-based approaches endows several benefits. Remarkably, 75-95% of relapses in lung cancer patients come with symptoms and, thus, a direct PRO measurement might be useful in the detection of an early disease progression. Easily accessible web-based application tools such as CANKADO were developed to report PROs more frequently compared to routine assessment. These tools help to strengthen the connection between patient and treating physician and to reduce patients' anxiety. Of note, even during treatment with toxic chemotherapy, most patients are willing and able to self-report via the web. Physicians appreciate PROs and trust in patient-reported information. In line with this, several promising studies confirmed a benefit from proactive, web-based monitoring programs. If symptoms occurred or worsened, the respective physician was informed earlier what resulted n improved OS, quality of life (QoL) and also in economic advantages due to less unnecessary routine check-ups. So far, these studies were performed on heterogeneous patient populations during chemotherapy. The current study is aimed to test the benefit of a web-based application tool in NSCLC, SCLC and TNBC patients during the recently approved first-line treatment strategy with atezolizumab in combination with chemotherapy.

ELIGIBILITY:
Inclusion criteria

1. Histologically or cytologically confirmed stage IV non-squamous NSCLC or histologically or cytologically confirmed extensive-stage SCLC or histologically or cytologically confirmed advanced (locally advanced and inoperable or metastatic), PD-L1 IC-positive TNBC, respectively
2. Indication and decision for approved therapy with

   1. atezolizumab and bevacizumab in combination with carboplatin and paclitaxel induction followed by atezolizumab/bevacizumab maintenance therapy in accordance with the current German SmPC of atezolizumab for first-line treatment of stage IV non-squamous NSCLC
   2. atezolizumab in combination with carboplatin and nab-paclitaxel induction followed by atezolizumab maintenance therapy in accordance to the current German SmPC of atezolizumab for first-line treatment of stage IV non-squamous NSCLC
   3. atezolizumab in combination with carboplatin and etoposide induction followed by atezolizumab maintenance therapy in accordance to the current German SmPC of atezolizumab for first-line treatment of extensive-stage SCLC
   4. atezolizumab in combination with nab-paclitaxel in accordance to the current German SmPC of atezolizumab for treatment of advanced, PD-L1 IC-positive TNBC
3. Aged ≥ 18 years
4. ECOG 0-2
5. In possession of a web-connected, frequently used, electronic device (smartphone, tablet, PC)
6. Willingness and ability to participate at the paper-based or digital questionnaire project and to participate at an initial training and to regularly use the web-based application tool CANKADO
7. Fluent in written and spoken German
8. Written (signed and dated) informed consent

Exclusion Criteria:

1. Prior treatment for stage IV non-squamous NSCLC (prior TKI therapy is allowed for EGFR mutant or ALK-positive NSCLC) or prior systemic treatment for extensive-stage SCLC or prior systemic chemotherapy for advanced TNBC
2. History of severe (or known) hypersensitivity to chimeric or humanized antibodies or fusion proteins or any component of atezolizumab formulation
3. Pregnant or breast-feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible are patients with histologically or cytologically confirmed stage IV NSCLC or extensive-stage SCLC who have already been scheduled to receive first-line treatment with atezolizumab in combination with platinum-based chemotherapy induction followed by atezolizumab-containing maintenance therapy according to the German SmPC (Fachinformation) OR patients with advanced (locally advanced and inoperable or metastatic), PD-L1 IC-positive TNBC who have been scheduled for first-line treatment with atezolizumab in combination with nab-paclitaxel according to the German SmPC (Fachinformation).
Sampling Method: Probability Sample
Enrollment: 154 (Actual)
Dates: Start 2019-07-10 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Overall Survival (OS) | 72 months
  Time from randomization to death from any cause. Patients not experiencing an event (i.e., patients alive at their individual end of study) will be censored with the last date the patient was known to be alive.

SECONDARY OUTCOMES:
Best response | 72 months
  The best documented response (in terms of complete response [CR], partial response [PR], stable disease [SD], or progressive disease [PD]) per patient, as assessed by the treating physician.
Overall response rate (ORR) | 72 months
  The proportion of patients showing a best overall response of CR or PR (as assessed by the treating physician).
Disease control rate (DCR) | 72 months
  The proportion of patients showing a best overall response of CR, PR, or SD (as assessed by the treating physician).
Progression Free Survival (PFS) | 72 months
  The time from randomization to tumor progression or death from any cause, whatever occurs first. Patients being event-free (i.e., alive and progression-free) by the time of analysis or starting a new antineoplastic therapy before progression, will be censored at the date of the last adequate tumor assessment.
Change from baseline in the global health scale score | 72 months
  To compare patient-reported outcomes (PROs) on quality of life (QoL) of the two study arms: Change from baseline in the global health scale score
Change from baseline in the functional/symptom scores | 72 months
  To compare patient-reported outcomes (PROs) on quality of life (QoL) of the two study arms: Change from baseline in the functional/symptom scores
Time to deterioration in global health scale score | 72 months
  To compare patient-reported outcomes (PROs) on quality of life (QoL) of the two study arms: Time to deterioration (TTD) by ≥ 10 points in the global health scale score
Time to deterioration in functional/symptom scores | 72 months
  To compare patient-reported outcomes (PROs) on quality of life (QoL) of the two study arms: Time to deterioration (TTD) by ≥ 10 points in the functional/symptom scores
Alerts | 72 months
  Frequency and total number of eHealth Support system (EHSS) alerts.
Sensitivity of alerts | 72 months
  Ratio of alert-initiated visits that result in detection of tumor progression and/or action-requiring symptom management (as evaluated by the oncologist) and all visits which result in detection of tumor progression and/or action-requiring symptom management.
Specifity of alerts | 72 months
  Ratio of non-alert-initiated visits with neither detected tumor progression nor action-requiring symptom management (as evaluated by the oncologist) and all visits with neither detected tumor progression nor action-requiring symptom management.
Positive predictive value of alerts | 72 months
  Ratio of alert-initiated visits that resulted in detection of tumor progression and/or action-requiring symptom management and all alert-initiated visits.
Negative predictive value of alerts | 72 months
  Ratio of non-alert-initiated visits with no result (i.e., neither detected tumor progression nor action-requiring symptom management) and all non-alert-initiated visits.
Progression-detection rate | 72 months
  The proportion of individuals who test positive for a first tumor progression during atezolizumab therapy in a specific type of tumor assessment (i.e., alert-triggered vs. non-alert-triggered), compared to the total number of first detected progressions during atezolizumab therapy (i.e., progressions detected in all tumor assessments during scheduled as well as unscheduled visits).
Patient compliance | 72 months
  Intensity of use of application tool (defined as number of utilizations per week over the total observation time).
Safety and tolerability | 72 months
  Frequency and severity of (serious) adverse events ((S)AEs) coded by the Medical Dictionary for Regulatory Activities (MedDRA), summarized by Preferred Term and System Organ Class and graded according to CTCAE v5.0.
  Frequency and severity of (serious) adverse drug reactions ((S)ADRs) with causal relationship to bevacizumab and/or atezolizumab coded by the MedDRA, summarized by Preferred Term and System Organ Class and graded according to CTCAE v5.0.
Treatment duration of first-line atezolizumab | 72 months
  Treatment duration of first-line atezolizumab (including maintenance therapy)
Relative dose intensity of first-line atezolizumab | 72 months
  Relative dose intensity of first-line atezolizumab (including maintenance therapy)
Treatment duration of each combined first-line antineoplastic therapy substance | 72 months
  Treatment duration of each combined first-line antineoplastic therapy substance
Relative dose intensity of each combined first-line antineoplastic therapy substance | 72 months
  Relative dose intensity of each combined first-line antineoplastic therapy substance
Treatment duration of combined first-line bevacizumab | 72 months
  Treatment duration of combined first-line bevacizumab (including maintenance therapy)
Treatment modifications of first-line atezolizumab and all combined antineoplastic substances | 72 months
  Therapy details and subsequent therapy lines based on Treatment modifications of first-line atezolizumab and all combined antineoplastic substances
Subsequent antineoplastic therapy lines | 72 months
  Therapy details and subsequent antineoplastic therapy lines
Subscale scores and single item responses | 72 months
  To compare patient-reported outcomes (PROs) on quality of life (QoL) of the two study arms Subscale scores and single item responses in Patient Reported Outcomes on QoL in both arms

CONTACTS AND LOCATIONS:
Overall Officials: Manfred Welslau, Dr., Principal Investigator — MVZ am Klinikum Aschaffenburg
Locations (92):
- Germany (92):
  - Onkologische Praxis im St. Marien-Krankenhaus, Ahaus
  - Gesundheitszentrum St. Marien, Amberg
  - Klinikum Arnsberg, Karolinen Hospital, Arnsberg
  - MVZ am Klinikum Aschaffenburg, Aschaffenburg
  - Klinikum Augsburg, II. Medizinische Klinik, Augsburg
  - Gemeinschaftspraxis Dr. Heinrich, Prof. Dr. Bangerter, Augsburg
  - Klinikum Bayreuth GmbH, Bayreuth
  - Facharztpraxis am VPH Bensberg, Onkologie und Hämatologie, Bergisch Gladbach
  - Onkologisches Versorgungszentrum Friedrichshain, Berlin
  - Praxiskooperation Bonn-Euskirchen, Bonn
  - Ev. Krankenhaus Göttingen-Weende gGmbH, Pneumologie, Beatmungsmedizin/Schlaflabor, Bovenden
  - Hämato- Onkologische Praxis im Medicum, Bremen
  - Klinikum Bremen-Ost, Pneumologie, Beatmungsmedizin, Bremen
  - MVZ am Allgemeinen Krankenhaus, Celle
  - MVZ des Städtischen Klinikums Dessau GmbH, Dessau
  - Onkologiezentrum Donauwörth, Donauwörth
  - Klinikum Dortmund, Pneumologie, Infektiologie, internistische Intensivmedizin, Dortmund
  - Onkologische Gemeinschaftspraxis, Dresden
  - Sana Kliniken Duisburg GmbH, Duisburg
  - Klinikum Esslingen GmbH, Esslingen am Neckar
  - Berufsausübungsgemeinschaft am Klinikum, Frankfurt (Oder)
  - Centrum für Hämatologie und Onkologie Bethanien, Frankfurt a.M.
  - Klinikum Frankfurt Höchst Innere Medizin 3, Frankfurt a.M.
  - Praxis Internistischer Onkologie und Hämatologie (PIOH), Frechen
  - Praxis für interdisziplinäre Onkologie & Hämatologie, Freiburg im Breisgau
  - Onkologische Schwerpunktpraxis, Freital
  - Gemeinschaftspraxis Panagiotou/Minaei (GbR), Garbsen
  - MVZ II der Niels Stensen Kliniken, Onkologie u. Hämatologie, Georgsmarienhütte
  - SRH Wald-Klinikum Gera GmbH, Gera
  - Universitätsklinikum Gießen, Medizinische Klinik V, Internistische Onkologie und Palliativmedizin, Giessen
  - Überörtliche Berufsausübungsgemeinschaft, Goslar
  - OSP Göttingen, Dres. Meyer / Ammon / Metz, Göttingen
  - Krankenhaus Martha-Maria Halle-Döla, Halle
  - Elbpneumologie im Struenseehaus, Hamburg
  - Evangelisches Krankenhaus Hamm gGmbH, Hamm
  - MediProjekt GbR, Hanover
  - DIAKOVERE Henriettenstift, Hanover
  - Westküstenkliniken Brunsbüttel und Heide, Medizinische Klinik I, Innere Medizin, Hämatologie, Onkologie, Heide
  - Onkologische Schwerpunktpraxis Dr. med. Volker Petersen, Heidenheim
  - Gemeinschaftskrankenhaus Herdecke, Herdecke
  - Frauenarztpraxis Dr. Lorenz, Hildburghausen
  - Praxisgemeinschaft Gynäkologische Onkologie & Spezielle Operative, Gynäkologie, Hildesheim
  - St. Bernward Krankenhaus, Hämatologie & Internistische Onkologie, Hildesheim
  - Onkologische Praxis, Hildesheim
  - Universitätsklinikum des Saarlandes, Homburg (Saar)
  - Gynäko-Onkologische Praxis, Ilsede
  - St. Vincentius-Kliniken gAG, Gynäkologie und Geburtshilfe, Karlsruhe
  - Hämato-Onkologisches Zentrum Kassel, Kassel
  - Internisten am Markt, Köthen
  - Zentrum für ambulante gynäkologische Onkologie - ZAGO, Krefeld
  - Onkologische Schwerpunktpraxis, Kronach
  - ÜBAG - MVZ Dr. Vehling-Kaiser GmbH Landshut, Landshut
  - POIS - Leipzig GbR Geßner u. Geßner, Leipzig
  - Onkologische Schwerpunktpraxis, Loerrach
  - Klinik Löwenstein, Löwenstein
  - Universitätsklinikum Gießen und Marburg, Marburg
  - Onkologische Gemeinschaftspraxis, Mayen
  - Gemeinschaftspraxis für Hämatologie und internistische Onkologie, Mülheim
  - Hämato-Onkologische Überörtliche Gemeinschaftspraxis, München
  - Thoraxzentrum Bezirk Unterfranken, Münnerstadt
  - Praxis Dr. med. Jens Uhlig, Naunhof
  - MVZ für Onkologie und Hämatologie im Rhein-Kreis Neuss, Neuss
  - MVZ Onko Medical GmbH Neustadt, Innere Med./Hämatologie-Onkologie, Neustadt am Rübenberge
  - Hämatologisch-Onkologische Gemeinschaftspraxis, Nordhorn
  - medius KLINIK NÜRTINGEN, Nürtingen
  - Onkologie Offenburg, Ambulantes Therapiezentrum für Hämatologie und Onkologie, Offenburg
  - Onkologische Praxis Oldenburg, Oldenburg
  - Pius-Hospital Oldenburg Universitätsklinik f. Innere Medizin Hämatologie und Onkologie, Oldenburg
  - Praxis Dagmar Guth, Plauen
  - Carl-von-Basedow-Klinikum, Medizinischen Klinik III, Pneumologie, Querfurt
  - Praxis für Hämatologie und internistische Onkologie, Ratingen
  - Praxis und Tagesklinik für Onkologie und Hämatologie, Recklinghausen
  - Onkologische Praxis Remscheid, Remscheid
  - Praxis und Tagesklinik für Onkologie und Hämatologie, Remscheid
  - Elblandkliniken Stiftung & Co. KG, Elblandklinikum Riesa, Riesa
  - Klinikum Südstadt Rostock, Innere Medizin III, Rostock
  - Zentrum für Urologie und Onkologie, Rostock
  - Praxis Dipl.-Med. René Schubert, Scheibenberg
  - Diakonie-Klinikum Schwäbisch Hall, Frauenklinik, Schwäbisch Hall
  - ZAHO Siegburg, Siegburg
  - MVZ Kloster Paradiese GbR, Soest
  - Hämatologie - Onkologie - Stolberg, Stolberg
  - g.SUND Gynäkologie Kompetenzzentrum Stralsund, Stralsund
  - Vinzenz von Paul Kliniken, Stuttgart
  - Praxisnetzwerk Hämatologie / internistische Onkologie, Troisdorf
  - SHG Kliniken Völklingen, Innere Medizin, Pneumologie, Thorakale Onkologie, Palliativmedizin, Völklingen
  - MVZ Weiden GmbH, Weiden
  - Gemeinschaftspraxis für Hämatologie und Onkologie, Westerstede
  - Praxisgemeinschaft für Onkologie und Urologie, Wilhelmshaven
  - GIM - Gemeinschaftspraxis Innere Medizin, Witten
  - MVZ West GmbH Würselen Hämatologie-Onkologie, Würselen
  - Praxis und Tagesklinik für Hämatologie/Onkologie, Zittau

IPD SHARING:
Plan to Share IPD: No